CLINICAL TRIAL: NCT01969487
Title: Effect of Preoperative Warmup on a Simulator by Trainee Surgeons on Intraoperative Robotic Surgical Skill and Postoperative Patient Outcomes
Brief Title: Effect of Preoperative Simulator Warmup on Intraoperative Robotic Surgical Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: NA_00074621; WU_00074621 (Other: Other)
Record Dates: First submitted 2013-09-25; First posted 2013-10-25 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Robotic Hysterectomy (Benign Indications/Early-stage Cancer)
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preoperative warm-up on simulator (Experimental): Trainees perform standard practice tasks programmed into a robotic surgical simulator immediately before the surgery.
  Interventions: Other: Preoperative warm-up on simulator
- No preoperative warm-up (No Intervention)

INTERVENTIONS:
Other: Preoperative warm-up on simulator
  Arms: Preoperative warm-up on simulator

SUMMARY:
Surgical residents and fellows acquire operative knowledge and skills by assisting attending surgeons in the operating room. Previous research has shown that practising technical skills prior to operating on patients can improve how skillfully laparoscopic surgery can be performed. Although an increasingly large number of patients are undergoing robotic hysterectomy and other robotic surgical procedures, little is known on how to ensure patient safety and treatment effectiveness when trainee surgeons participate in the operating room. Our study aims to determine the impact of immediate preoperative warm-up on a robotic surgery simulator by gynecologic surgical trainees on their intraoperative performance and on patient outcomes. The investigators are randomly assigning gynecologic surgical trainees at a major academic medical center to either warm-up immediately before surgery on a robotic surgery simulator or to not warm-up. The attending surgeon supervising the trainee in the operating room is unaware of whether the trainee was assigned to warm-up or no warm-up. The investigators will compare standard robotic surgical skills assessments of the trainees by the supervising attending surgeons and patient outcomes in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the graduate (residency and fellowships) gynecology training program at the study institution;
* Participation as assistant surgeon in a robotic hysterectomy for benign indications for early stage uterine or cervical cancer.

Exclusion Criteria:

* Participation as assistant surgeon in a non-robotic hysterectomy or robotic hysterectomy for gynecologic cancer that has spread beyond the uterus based on preoperative imaging and biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Global rating score - GEARS approach | Assessed during the surgery (scheduled immediately following warm-up/no warm-up)
  Global rating scores assigned by the supervising surgeon immediately after each study surgical procedure. Global rating scores use two different approaches - the Objective Structured Assessment of Surgical Skills (OSATS) and the Global Evaluative Assessment of Robotic Surgery (GEARS).
Global rating score - OSATS approach | Assessed during the surgery (scheduled immediately following warm-up/no warm-up)
  Global rating scores assigned by the supervising surgeon immediately after each study surgical procedure. Global rating scores use two different approaches - the Objective Structured Assessment of Surgical Skills and the Global Evaluative Assessment of Robotic Surgery.
Surgical skill metrics | Assessed during the surgery (scheduled immediately following warm-up/no warm-up)
  Computed using surgical tool motion and/or video of procedure.

SECONDARY OUTCOMES:
Operative time | Intraoperative
Estimated blood loss | Intraoperative
Length of hospital stay | We will follow patients in the study for the duration of their hospital stay; an anticipated average of about 5 days.
Change in hematocrit | Postoperative days 1, 2, and 3
Readmission or emergency room visit | 6 weeks after discharge from hospital (following initial admission for surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Grace CC Chen, M.D., Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland